CLINICAL TRIAL: NCT01002677
Title: Midwest Advocacy Project: A Community-based Randomized Practical Behavioral Trial of Programmed Advocacy Training for Individuals With Traumatic Brain Injury and Their Significant Others
Brief Title: Behavioral Trial Studying Programmed Training to Improve Advocacy Skills for Individuals With Traumatic Brain Injury
Acronym: MAP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Allen Brown, Director, Brain Rehabilitation Research, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 08-000981; H133A070013-09
Record Dates: First submitted 2009-10-22; First posted 2009-10-27 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Brain Injuries
Keywords: brain injury; traumatic brain injury; training; teaching; curriculum
MeSH Terms: conditions — Brain Injuries; Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Curriculum (Experimental)
  Interventions: Behavioral: Advocacy training curriculum
- Self-directed (Active Comparator)
  Interventions: Behavioral: Self-directed

INTERVENTIONS:
Behavioral: Advocacy training curriculum — Day-long presentation of an advocacy training curriculum by the state's Brain Injury Association staff: One session per month for 4 consecutive months.
  Arms: Curriculum
Behavioral: Self-directed — Day-long group-based self-directed advocacy training activity: One session per month for 4 consecutive months.
  Arms: Self-directed

SUMMARY:
The Midwest Advocacy Project (MAP) is a community-based multiple-site randomized practical behavioral trial of advocacy skill training for individuals with traumatic brain injury (TBI), their families, and significant others. The purpose is to evaluate the efficacy of a 4-session advocacy training program to improve behavioral advocacy skills compared to self-directed advocacy training of the same session frequency. Groups will be randomly assigned to either a programmed group or a self-directed group in collaboration with the Brain Injury Associations of Minnesota, Iowa, and Wisconsin each year over the 5 year study period. The primary outcome is pre-post measures of written and verbal advocacy skill measured by the Advocacy Behavior Rating Scale.

It is hypothesized that subjects who receive programmed advocacy training will show greater positive change on pre-post measures of advocacy skill measures than subjects receiving self-directed training.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* moderate-severe TBI as indicated by one of the following:
* post traumatic amnesia (PTA) > 24 hours
* or loss of consciousness > 30 minutes
* or neuroimaging evidence of trauma-related intracranial abnormality
* Or the family/significant other of an individual with TBI meeting the above criteria
* 1 or more years post-injury
* Functional English speaker
* Signed consent to participate

Exclusion Criteria:

* Severe cognitive impairment as indicated by one or more of the following:
* Disorientation to person or year
* Unable to complete pre-program interview because of severe communication limitations
* Unable to remember important information given in the course of the pre-program interview, such as, time and place of program, number of sessions, and contact person
* Unable to complete the pre-program interview because of loss of emotional control, such as, extended tearfulness, sustained anger, verbal attack on interviewer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2007-08; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Score on the Advocacy Behavior Rating Scale | Written and verbal (video) advocacy statements are obtained twice from each subject and rated by blinded investigators: once after consenting and before beginning the group's advocacy activity, and; after the last advocacy activity session 4 weeks later.

SECONDARY OUTCOMES:
Score on Advocacy Activity Scale | The Advocacy Activity Scale score is obtained twice from each subject: once after consenting and before beginning the group's advocacy activity, and; after the last advocacy activity session 4 weeks later.
Score on the Perceived Control Scale for Brain Injury | The Perceived Control Scale for Brain Injury score is obtained twice from each subject: once after consenting and before beginning the group's advocacy activity, and; after the last advocacy activity session 4 weeks later.
The Craig Hospital Inventory of Environmental Factors-Short Form | The Craig Hospital Inventory of Environmental Factors-Short Form score is obtained twice from each subject: once after consenting and before beginning the group's advocacy activity, and; after the last advocacy activity session 4 weeks later.
The Satisfaction with Life Scale | The Satisfaction with Life Scale is obtained twice from each subject: once after consenting and before beginning the group's advocacy activity, and; after the last advocacy activity session 4 weeks later.
The SF-12 | The SF-12 score is obtained twice from each subject: once after consenting and before beginning the group's advocacy activity, and; after the last advocacy activity session 4 weeks later.
Advocacy Activity Scale | Every 6 months after intervention until the end of the 5-year study period

CONTACTS AND LOCATIONS:
Overall Officials: Allen W Brown, MD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Brain Injury Association of Iowa, Urbandale, Iowa
  - Brain Injury Association of Minnesota, Minneapolis, Minnesota
  - Brain Injury Association of Wisconsin, Pewaukee, Wisconsin